CLINICAL TRIAL: NCT02674971
Title: Lowering Caloric Density of the Diet
Acronym: Lower CD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UTKIRB-15-02609
Record Dates: First submitted 2016-01-25; First posted 2016-02-05 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Feeding Behavior
MeSH Terms: conditions — Obesity; Feeding Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- INCREASE (Active Comparator): This condition will be instructed to make food consumption decisions based solely upon the ED of a food. The goal of the ED condition will be to consume at least 10 foods ≤ 1.0 kcal/g (i.e., fruits and vegetables, broth based soups, non-fat yogurts, some legumes, egg substitutes, some white fish, etc.) per day.
  Interventions: Behavioral: Common components of intervention
- COMBINATION (Active Comparator): This condition will be identical to the INCREASE condition, except it will also have a goal regarding the number of high-ED foods to consume and substituting low-ED foods for high-ED foods. Thus, this condition will have ED goals to consume at least 10 foods ≤ 1.0 kcal/g (i.e., fruits and vegetables, broth based soups, non-fat yogurts, some legumes, egg substitutes, some white fish, etc.) and no more than 2 foods ≥ 3.0 kcal/g (i.e., crackers, chips, cookies, hard cheeses, hot dogs, salad dressings, etc.) per day. Foods with an ED >1.0 kcal/g but < 3.0 kcal/g will be unlimited; however, lower ED foods will be strongly encouraged. Furthermore, additions to beverages (i.e., sugar, cream) will count toward the > 3.0 kcal/g goal if the additions meet that ED criteria.
  Interventions: Behavioral: Common components of intervention

INTERVENTIONS:
Behavioral: Common components of intervention — 12-week standard lifestyle intervention for obesity, which consists of weekly meetings. Each meeting will last 60 minutes, with participants attending group meetings specific for their condition. In all meetings, participants will be weighed, homework assignments will be verbally reviewed, and a behavioral lesson will be presented. Basic behavioral lessons, will be similar to those that have been successfully used in the Diabetes Prevention Program (DPP) and Look AHEAD. Topics to be covered in the meetings will focus on the dietary prescriptions and dietary information for each condition, the physical activity goal, energy balance, and behavioral strategies. Each session will conclude with reminding participants of their dietary and physical activity goals, and having participants self-monitor these behaviors every day and implement the behavioral strategies discussed in the session.

SUMMARY:
For weight loss to occur, energy intake needs to be reduced to incur an energy deficit. One dietary strategy that may facilitate reducing energy intake and enhancing weight loss is consuming a diet low in dietary energy density (ED). The ED of a given food, defined as the ratio of energy of the food to the weight of the food (kcal/g), is largely determined by water content, but is also affected by fat and fiber. Although the 2010 Dietary Guidelines encourage an eating pattern low in energy density (ED) to manage weight, it is currently not known what the best strategy is for reducing ED in the diet. Eating a greater number of foods low in ED or reducing the number of foods high in ED may reduce overall dietary ED. As ED is believed to reduce intake by allowing a greater weight of food relative to total energy consumed assisting with enhancing feelings of fullness, it is anticipated that either increasing consumption of low-ED foods in the diet alone or combining an increase in consumption of low-ED foods with a decrease in consumption of high-ED foods may be the best strategies for reducing overall dietary ED for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* 1) age between 18 and 65 years and 2) a body mass index (BMI)7 between 27 and 45 kg/m2.

Exclusion Criteria:

1. report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q)8 (medical conditions that could limit exercise for safety reasons will be required to obtain written physician consent before participating in the investigation)
2. report being unable to walk for 2 blocks (1/4 mile) without stopping
3. are currently participating in a weight loss program and/or taking weight loss medication or lost > 5% of body weight during the past 6 months
4. report major psychiatric diseases or organic brain syndromes
5. have had bariatric surgery or are planning to have bariatric surgery within the next 4 months
6. intend to move outside of the metropolitan area within the time frame of the investigation
7. are pregnant, lactating, < 6 months post-partum, or plan to become pregnant during the investigation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dietary: Energy Intake | change from baseline to 12 weeks
  Changes in overall dietary intake and changes per eating bout will be assessed by 3 day (2 weekdays and 1 weekend) food records. To determine dietary variables, each food record will be entered into the Nutrition Data System for Research (NDS-R) software developed by the Nutrition Coordinating Center, University of Minnesota, Minneapolis, Minnesota.
Physical activity | change from baseline to 12 weeks
  Changes in self-reported physical activity will be determined by the Paffenbarger Activity Questionnaire (PAQ).16 This questionnaire yields estimates of the total energy expended in PA per week based on flights of stairs climbed per day, city blocks walked per day, and hours of structured activity acquired within a typical week. The PAQ has been shown to be significantly correlated with an objective measure of PA.
Ecological Momentary Assessment (EMA) | change from baseline to 12 weeks
  (EMA) refers to a collection of methods often used in behavioral medicine research by which a research participant repeatedly reports on symptoms, affect, behavior, and cognitions close in time to experience and in the participants' natural environment. EMA protocol will be conducted over 7 continuous days using both semi-random and event-contingent sampling. Semi-random responses will be collected at varied times within three windows (morning, afternoon, and evening), with three assessments occurring per day triggered by an alarm prompt that signals a 30-minute window for response. Event-based sampling will be used to assess eating bouts. Semi-random sampling will assess consumption cues (i.e. feelings of temptation, fullness, desire to eat, energy level and control over eating), along with feelings of hunger, satiation, and deprivation using a series of 11 questions.
Weight | change from baseline to 12 weeks
  Change in weight will be assessed by an electronic scale, using standard procedures.
Dietary: Grams of Intake | change from baseline to 12 weeks
  Changes in overall dietary intake and changes per eating bout will be assessed by 3 day (2 weekdays and 1 weekend) food records. To determine dietary variables, each food record will be entered into the Nutrition Data System for Research (NDS-R) software developed by the Nutrition Coordinating Center, University of Minnesota, Minneapolis, Minnesota.
Dietary: Energy Density | change from baseline to 12 weeks
  Changes in overall dietary intake and changes per eating bout will be assessed by 3 day (2 weekdays and 1 weekend) food records. To determine dietary variables, each food record will be entered into the Nutrition Data System for Research (NDS-R) software developed by the Nutrition Coordinating Center, University of Minnesota, Minneapolis, Minnesota.
Dietary: Macronutrients | change from baseline to 12 weeks
  Changes in overall dietary intake and changes per eating bout will be assessed by 3 day (2 weekdays and 1 weekend) food records. To determine dietary variables, each food record will be entered into the Nutrition Data System for Research (NDS-R) software developed by the Nutrition Coordinating Center, University of Minnesota, Minneapolis, Minnesota.
Dietary: Fiber | change from baseline to 12 weeks
  Changes in overall dietary intake and changes per eating bout will be assessed by 3 day (2 weekdays and 1 weekend) food records. To determine dietary variables, each food record will be entered into the Nutrition Data System for Research (NDS-R) software developed by the Nutrition Coordinating Center, University of Minnesota, Minneapolis, Minnesota.
Height | baseline
  Height will be assessed by stadiometer, using standard procedures.
BMI | change from baseline to 12 weeks
  Change in BMI (kg/m2) will be calculated from height and weight measures.

SECONDARY OUTCOMES:
Diet satisfaction | 12 weeks
  The Food Acceptability Questionnaires will assess acceptability and satisfaction of diet at 12 weeks. Participants will be asked about ease of following the diet, ease of determining foods to consume to meet dietary goals, and ease of reading food labels to select foods to consume to meet dietary goals (which is all one questionnaire).

OTHER OUTCOMES:
Demographic characteristics | baseline
Compliance | 12 weeks
  Participation will be recorded.
Weight History | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee, United States